CLINICAL TRIAL: NCT04892173
Title: A Phase 3 Study of NBTXR3 Activated by Investigator's Choice of Radiotherapy Alone or Radiotherapy in Combination With Cetuximab for Platinum-based Chemotherapy-Ineligible Elderly Patients With LA-HNSCC
Brief Title: JNJ-90301900 (NBTXR3) Activated by Radiotherapy With or Without Cetuximab in LA-HNSCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NANORAY-312; NANORAY-312 (Other: Janssen Research & Development, LLC); 2024-520386-31-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma; Aged
Keywords: LA-HNSCC; NBTXR3; hafnium oxide; radioenhancer; Radiotherapy; RT; HNSCC; radiation therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): JNJ-90301900 (NBTXR3), as an intratumoral/intranodal injection, activated by investigator's choice of RT alone or RT in combination with cetuximab. JNJ-90301900 (NBTXR3) is given as a dose of 33% of the Gross Tumor Volume.
  Interventions: Drug: JNJ-90301900 (NBTXR3); Drug: Cetuximab; Radiation: Radiation Therapy
- Arm B (Active Comparator): Investigator's choice of RT alone or RT in combination with cetuximab.
  Interventions: Drug: Cetuximab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: JNJ-90301900 (NBTXR3) — Suspension of inert, crystalline hafnium oxide particles, designed to generate oxygen free radicals to destroy cancer cells after activation by ionizing radiation.
  Other Names: Functionalized hafnium oxide nanoparticles; NBTXR3
  Arms: Arm A
Drug: Cetuximab — Solution for infusion
  Other Names: Erbitux
Radiation: Radiation Therapy — Intensity-modulated radiation therapy (IMRT): 70 Gray in 35 fractions over a 7-week period.

SUMMARY:
This is a global, open-label, randomized, 2-arm, Investigator's choice Phase 3 (Pivotal Stage) study to investigate the efficacy and safety of JNJ-90301900 (NBTXR3) / radiation therapy (RT)±cetuximab versus RT±cetuximab in treatment-naïve, platinum-ineligible, elderly participants with locally advanced head and neck squamous cell carcinoma (LA-HNSCC).

DETAILED DESCRIPTION:
Participants will undergo a screening assessment over a period of less than or equal to (<=) 28 days to determine eligibility.

Eligible participants will be treated by the Investigator's choice of RT alone or RT in combination with cetuximab. Following the Investigator's choice, participants will be randomized in a 1:1 ratio:

* Arm A: JNJ-90301900 (NBTXR3), as an intratumoral/intranodal injection, activated by investigator's choice of RT alone or RT in combination with cetuximab
* Arm B: Investigator's choice of RT alone or RT in combination with cetuximab

All participants (Arm A and Arm B) will receive 70 Gy in 35 fractions over a 7 week period.

An EOT visit will be performed 4 weeks after the completion of RT. Follow-up visits will start at 12 weeks post-RT completion, and will continue every 12 weeks for 2 years, and then every 24 weeks thereafter until death; the participant is determined to be lost to follow up; withdrawal of consent; or the end of the study, whichever occurs first. Participants who have received further anti-cancer therapy for the study disease and/or have had disease progression/recurrence will be followed only for survival information

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=) 60 years old
* Squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or supraglottic larynx and a candidate for definitive radiation therapy with or without cetuximab
* Clinical stage T3-4 NX or T2 N2-3 disease according to the 8th edition of AJCC
* One primary tumor lesion amendable for intratumoral injection
* Ineligible to receive platinum-based chemotherapy with radiation (at least one of the following):

  1. Estimated creatinine clearance >= 30 and less than (<) 50 milliliters/minute (mL/min) (per Cockcroft-Gault equation), Grade >= 2 hearing loss or tinnitus, Grade >= 2 peripheral neuropathy, Eastern Cooperative Oncology Group (ECOG) Performance Status 2 or New York Heart Association Class 3
  2. Age 70-74 years old with Geriatric 8 (G8) score less than or equal to (<=) 14
  3. Age >= 75 years old

Exclusion Criteria:

* Carcinoma of the nasopharynx, paranasal sinus(es), salivary gland, thyroid gland, or unknown primary
* Non-squamous cell histology
* Clinical stage T1-2 N0, T2 N1, or M1 disease according to the 8th edition of AJCC
* Loco-regionally recurrent head & neck cancer that has been previously treated with surgery, radiation therapy, and/or chemotherapy
* Prior or concurrent primary malignancy (including second synchronous head & neck cancer) within the last 2 years of informed consent and whose natural history has the potential to interfere with the safety and efficacy assessment of the investigational agent
* Ongoing or active infection requiring treatment with antimicrobial therapy within 2 weeks of randomization

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 30 months following first randomized participant
  Time from randomization to local-regional recurrence, local-regional progression, distant progression, or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | 48 months following first randomized participant
  Time from randomization to death from any cause
Local-regional control | 48 months following first randomized participant
  Time to local regional progression: time from Randomization to local-regional progression or death, whichever occurs first
Distant control | 48 months following first randomized participant
  Time to distant progression: time from Randomization to distant progression or death, whichever occurs first
Objective Response Rate (ORR) | 48 months following first randomized participant
  Rate of complete response (CR)+partial response (PR) [RESIST 1.1]
Duration of Overall Response | 48 months following first randomized participant
  Time from CR or PR to progression of disease, unequivocal clinical progression, or death, whichever occurs first
Quality of Life over time - QLQ H&N35 | 48 months following first randomized participant
  Change from baseline over time in symptoms, function, and health related QOL using the European Organisation for Research and Treatment of Cancer (EORTC) questionnaire-Head and Neck Cancer Module (QLQ H&N35)
Quality of Life over time - EQ 5D 5L | 48 months following first randomized participant
  Change from baseline over time in symptoms, function, and health related QOL using the 5 level EuroQol 5 dimension (EQ 5D 5L) instrument
Safety across duration of study - AEs | 48 months following first randomized participant
  Adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation Inc Clinical trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (188):
- United States (25):
  - City of Hope, Duarte, California
  - University of California at San Diego Moores Cancer Center, La Jolla, California
  - Memorial Radiation Oncology Medical Group Laguna Hills, Laguna Hills, California
  - UCLA Hematology Oncology, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - University of California San Francisco, San Francisco, California
  - George Washington University Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Richmond University Medical Center, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Macon Joan Brock Virginia Health Sciences Eastern Virginia Medical Group at Old Dominion University, Norfolk, Virginia
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Medizinische Universitaet Wien, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital De Charleroi Site Les Viviers, Charleroi
  - Universitair Ziekenhuis Leuven, Leuven
- Brazil (16):
  - Fundacao Pio Xii - Hospital De Cancer De Barretos, Barretos
  - Nucleo de Ensino e Pesquisa do Instituto Mario Penna, Belo Horizonte
  - Centro Regional Integrado de Oncologia CRIO, Fortaleza
  - Hospital Haroldo Juaçaba - Instituto do Câncer do Ceará, Fortaleza
  - Fundacao Sao Francisco Xavier, Ipatinga
  - Hospital Amaral Carvalho, Jaú
  - Hospital do Cancer de Londrina, Londrina
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Grupo Oncoclinicas - Botafogo, Rio de Janeiro
  - Ensino e Terapia de Inovacao Clinica AMO Etica, Salvador
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Hospital Sirio Libanes Sao Paulo, São Paulo
  - Associacao Feminina de Educacao e Combate ao Cancer Hospital Santa Rita de Cassia, Vitória
- Bulgaria (2):
  - MHAT Uni Hospital, Panagyurishte
  - Specialized Hospital for Active Treatment in Oncology, Sofia
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada
- China (35):
  - The Affiliated Hospital of Bengbu Medical College, Bengbu
  - Xiangya Hospital Central South University, Changsha
  - Hunan Cancer hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Dongguan People s Hospital, Dongguan
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Fujian Medical University Fujian Provincial Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou
  - Guangzhou Medical University Affiliated Oncology Hospital, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Cancer Hospital, Jinan
  - Linyi Cancer Hospital, Linyi
  - Liuzhou people's Hospital, Liuchow
  - Jiangxi Cancer Hospital, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Wuming Hospital of Guangxi Medical University, Nanning
  - The Cancer Hospital Affiliated to Guangxi Medical University, Nanning
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Second Affiliated Hospital, SooChow University, Suzhou
  - Shanxi Provincial Cancer hospital, Taiyuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The first affiliated hospital of xiamen university, Xiamen
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The Fifth Affiliated Hospital Sun Yat Sen University, Zhuhai
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice Bulovka, Prague
- Tampereen Yliopistollinen Sairaala, Tampere, Finland
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU Brest, Brest
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Centre de Lutte contre le Cancer Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Curie, Paris
  - Hopital Tenon, Paris
  - Hopital Haut Leveque, Pessac
  - Hopital Pontchaillou, Rennes
  - CLCC - Centre Henri Becquerel, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Centre Hospitalier de Valenciennes Hopital Jean Bernard, Valenciennes
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Georgia (4):
  - High Technology Hospital MedCenter Ltd Batumi, Batumi
  - JSC Vian Kutaisi Referral Hospital, Kutaisi
  - Todua Clinic, Tbilisi
  - Ltd Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
- Germany (5):
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Jena, Jena
  - Klinikum rechts der Isar an der Technischen Universitat Munchen, München
  - Universitaetsmedizin Rostock, Rostock
- Greece (4):
  - General Hospital of Athens Attikon, Athens
  - University Hospital Of Larissa, Larissa
  - Athens Medical Center S A Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Hungary (3):
  - Eszak Pesti Centrumkorhaz Honvedkorhaz, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Szent Gyorgyi Albert Klinikai Kozpont Onkoterapias Klinika, Szeged
- India (6):
  - M S Ramaiah Memorial Hospital, Bangalore
  - Apollo Speciality Hospital, Chennai, Chennai
  - Meenakshi Mission Hospital and Research Center, Madurai
  - Tata Memorial Hospital, Mumbai
  - HealthCare Global HCG Manavata Cancer Centre, Nashik
  - Grant Medical foundation Ruby Hall Clinic, Pune
- Israel (4):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (10):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Hiroshima University Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa
  - Aichi Cancer Center, Nagoya
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka Sayama Shi
  - Tohoku University Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke
  - Tokyo Medical University Hospital, Shinjuku
  - Shizuoka Cancer Center, Sunto Gun
- Philippines (4):
  - University of Perpetual Help Dalta Medical Center, Inc, Las Piñas
  - Manila Doctors Hospital, Manila
  - The Medical City, Pasig
  - St. Luke's Medical Center, Quezon City
- Portugal (5):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Hosp. Cuf Descobertas, Lisbon
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Uls Gaia Espinho, Vila Nova de Gaia
- Institutul Oncologic Prof Dr Al Trestioreanu Bucuresti, Bucharest, Romania
- Serbia (4):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Vojnomedicinska Akademija, Belgrade
  - Institute of Oncology of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
- South Korea (4):
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Asan Medical Center (AMC), Seoul
  - The Catholic university of Korea, St. Vincent's Hospital, Suwon
- Spain (17):
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Instituto Catalan Deoncologia Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospitales Universitarios San Roque En Las Palmas de Gran Canaria Centro Oncologico Integral Canario, Las Palmas de Gran Canaria
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. de Navarra, Pamplona
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Inst. Valenciano de Oncologia, Valencia
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Taiwan (5):
  - National Cheng Kung University Hospital, Bei Qu
  - Changhua Christian Hospital, Changhua
  - Chang-Gung Memorial Hospital-Keelung, Keelung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - The Royal Marsden NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Tourneau C, Takacsi-Nagy Z, Nuyts S, Thureau S, Liu F, Hoffmann C, Hackman TG, Lesnik M, Debard A, Finzi L, Devisetty K, Vivar OI, Farber LA, Nguyen F, Liem X, Natelauri E, Psyrri A, Burian M, Yu J, Yom SS. Nanoray-312: phase III study of NBTXR3 + radiotherapy +/- cetuximab in elderly, platinum-ineligible locally advanced HNSCC. Future Oncol. 2025 May;21(12):1489-1499. doi: 10.1080/14796694.2025.2496131. Epub 2025 May 5. PMID 40323213